CLINICAL TRIAL: NCT05370651
Title: A Single-Blind, Randomized Study of the BTL Emsella Chair Versus Sham for the Treatment of Male Sexual Dysfunction
Brief Title: Emsella Chair vs Sham for Male Sexual Dysfunction
Acronym: Emsella_EJD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Director and Chair of the Department of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-165
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Male Sexual Dysfunction; Ejaculatory Dysfunction
Keywords: Male Sexual Dysfunction
MeSH Terms: conditions — Ejaculatory Dysfunction

STUDY DESIGN:
Intervention Model Description: We will be performing this study in 2 phases: Phase 1 will be an open label pilot study of 10 male participants. All participants in the pilot study will receive active treatment. If data from the pilot study is suggestive of symptom improvement, we will continue enrolling participants on to phase 2, which is a sham controlled, randomized blinded study. Patients who meet all eligibility criteria will be randomized (2:1) to receive Emsella chair or sham treatments. In phase 2, the subject and biostatistician will be blinded to the group allocation throughout the study. The initial analysis of data, performed by the biostatistician will not include group assignment.
Who Masked: Participant, Outcomes Assessor
Masking Description: The sham Emsella treatment will provide sensation without active HIFEM technology. The sham treatment amplitude setting will be limited to below the therapeutic level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Emsella Chair Active Treatment (Active Comparator): Subjects will be asked to sit on the device and the height will be adjusted until the subject's feet are on the floor. The active treatments are individualized, since some subjects will be more sensitive than others. The Emsella chair will be turned on and the setting gradually increased to the subject's sensory threshold; the maximum sensation the subject can tolerate. The setting will be decreased slightly and stay unchanged for the remainder of the treatment. The treatment threshold should be increased with every treatment until the subject reaches 100%.
  Interventions: Device: BTL Emsella Chair
- Emsella Chair Sham Treatment (Sham Comparator): Sham treatment subjects will be positioned on the device in the same manner. The sham treatment will provide some sensation without active HIFEM technology. The programming for the sham treatment will have an amplitude limitation, with the setting below the therapeutic level (<10% power).
  Interventions: Device: BTL Emsella Chair

INTERVENTIONS:
Device: BTL Emsella Chair — Subjects will sit on the device. The clinical research coordinator will turn the device on and increase the setting gradually until the patient reaches their sensory threshold. This is the maximum sensation the patient can tolerate. The treatment threshold should be increased until the subject reaches 100%.

SUMMARY:
We will be performing this study in 2 phases: Phase 1 will be an open label pilot study of 10 male participants. All participants in the pilot study will receive active treatment. If data from the pilot study is suggestive of symptom improvement, we will continue on to phase 2, which is a sham controlled, randomized blinded study. Participants in phase 2 will be randomized to receive either active treatment or sham. Potentially a total of 117 participants for both phases will be enrolled.

The purpose of this study is to compare the Emsella Chair to sham and to determine whether electromagnetic technology is effective in the treatment of sexual dysfunction, specifically erectile dysfunction (EjD) in men.

DETAILED DESCRIPTION:
Male sexual health is an often overlooked and ignored facet of mens well-being. However, this can have significant effects on quality of life for both the man afflicted by sexual dysfunction as well as their partner. Most commonly we think of erectile dysfunction (ED) as the main factor of male sexual dysfunction, but ejaculatory dysfunction (EjD) and other problems relating to orgasm are also important. EjD is exceedingly common especially in the aging male population, and includes premature ejaculation (PE), delayed ejaculation (DE), anejaculation (absence of ejaculation during orgasm), retrograde ejaculation, and painful ejaculation. Medications such as sildenafil (Viagra) and tadalafil (Cialis) are Phosphodiesterase type 5 (PDE-5) inhibitors that are commonly used for the treatment of ED, but there are very few medications specifically formulated to treat EjD. More conservative management options for the treatment of ED include vacuum erection devices, psychotherapy, and lifestyle changes. The usual next step after failure of the above options includes intracavernosal injections which involve directly injecting erectogenic medication into the penis, intraurethral injections, or finally surgery. Ejaculatory dysfunction on the other hand, whether it be premature, delayed, retrograde, or anejaculation all have much less treatment options. Most of these include either the off-label use of medications to treat other conditions or sex therapy / psychotherapy.

Treatments including pudendal neuromodulation or pudendal canal decompression have shown significant improvement in ED and EjD. Due to side effects and the lack of patient compliance to oral medication, non-oral medication treatments are in high demand for this condition. Neuromodulation therapies have become increasingly popular for the treatment of male sexual dysfunction. These neuromodulation therapies often work by stimulating the sacral nerve. The Emsella Chair is a conservative neuromodulation therapy that may have a role for patients who are not surgical candidates or who desire a noninvasive treatment option. The Emsella Chair uses high intensity focused electromagnetic (HIFEM) technology to induce deep pelvic floor muscle contractions, the equivalent of 11,200 Kegel exercises over 28 minutes. The treatment awakens deconditioned pelvic floor muscles, delivers the stimulations, and then relaxes the muscles. The repetition of these phases leads to pelvic floor adaptation and remodulation. this treatment could provide similar improvement for men with sexual dysfunction given the significant overlap in anatomy and physiology, as well as studies that have shown improvement in sexual dysfunction with pelvic floor muscle therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and provide written, dated, informed consent prior to screening, and be likely to comply with study protocol, including independently complete study questionnaires and communicate with study personnel about adverse events and other clinically important information.
2. Men ≥ 18 years of age.
3. Sexually active within the past 12 weeks and plan to be sexually active during the next 12 weeks.

5. Self-reported ejaculatory dysfunction symptoms present >3 months 6. Self-reported failed conservative care of behavioral modifications and/or oral medications.

7. Subject agrees not to start any new treatment for erectile dysfunction or ejaculatory dysfunction during the treatment and follow-up periods.

Exclusion Criteria:

1. Botox® use in bladder or pelvic floor muscles in the past year
2. Subject weighs greater than 330 pounds, due to weight limits of the Emsella Chair.
3. Pulmonary insufficiency, defined as difficulty breathing and fatigue, especially during exercise; chest pain, such as squeezing, pressure of tightness; the sensation of rapid or irregular heartbeat (palpitations); swelling of the legs or feet; dizziness or fainting; and/or bluish discoloration of the nails and/or lips (cyanosis)
4. Any condition that causes a lack of normal skin sensation to the pelvis, thigh, or buttocks.
5. Major metal implants such as: metal plates, screws, joint replacements, implanted cardiac pacemakers, drug pumps, neurostimulators, electronic implants, defibrillators, and metal implants in the pelvic area. Patients with other metal implants will be evaluated by the investigator for inclusion in the study.
6. Previous or current penile prosthesis.
7. Subject has a piercing between the waist and knees and is not willing to remove it before each treatment
8. Active urethral diverticula
9. Known history of urethral stricture disease
10. Currently healing from surgical procedures where muscle contraction may disrupt the healing process
11. Subject is currently receiving treatment for a malignant tumor that would interfere with study participation.
12. Subject has used the BTL EMSELLA device previously
13. Subject has sexual dysfunction of neurogenic etiology, such as multiple sclerosis, spina bifida, Parkinson's, spinal cord injury, diabetic neuropathy, neurogenic bladder etc.
14. Current use of neuromodulation therapy, including Interstim and percutaneous tibial nerve stimulation (PTNS), for bladder symptoms within 3 months of screening visit (if past sacral/pudendal implant, must be explanted)
15. Currently participating in an investigational study that may impact study results or previously received an investigational drug or treatment within 30 days of the Screening Visit
16. Current or history of any physical condition that, in the investigator's opinion, might put the subject at risk or interfere with study results interpretation

    * Note for the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must a male, with male genitals
Enrollment: 117 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The overall efficacy of the Emsella Chair to sham by evaluating subject reported symptom improvement as measured by the Global Response Assessment (GRA) | 4 weeks after completing all 8 treatments
  The GRA is a validated single question survey prompting subjects to rank change in symptom severity since the start of therapy on a 7-point scale (1 = markedly worse, 2 = moderately worse, 3 = mildly worse, 4 = same, 5= slightly improved, 6 = moderately improved, 7= markedly improved). A score equal to or above 5 will show improvement. A score of 4 will mean no change. A score equal to or below 3 will show worsening of symptoms.

SECONDARY OUTCOMES:
Change in subject-reported ability to achieve an erection as measured by the Male Sexual Health Questionnaire (MSHQ) responses. | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score for Question 1 will be reviewed from the erection scale. "In the last month, without using drugs like Viagra, how often have you been able to get an erection when you wanted to?" Measured as (5 = all of the time, 4 = most of the time, 3 = about half of the time, 2 = less than half the time, 1 = none of the time, and 0= used Viagra or similar drug with every sexual encounter). A higher score indicates a higher ability to achieve an erection. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported ability to maintain an erection as measured by MSHQ responses | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 2 will be reviewed from the erection scale. "In the last month, if you were able to get an erection without using drugs like Viagra, how often were you able to stay hard as long as you wanted to?" Measured as (5 = all of the time, 4 = most of the time, 3 = about half of the time, 2 = less than half the time, 1 = none of the time, and 0= used Viagra or similar drug with every sexual encounter). A higher score indicates a higher ability to maintain an erection. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported ability to ejaculate as measured by MSHQ responses | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 5 will be reviewed from the ejaculation scale. "In the last month, how often have you been able to ejaculate when having sexual activity?" Measured as (5 = all of the time, 4 = most of the time, 3 = about half of the time, 2 = less than half the time, 1 = none of the time/could not ejaculate). A higher score indicates a higher ability to achieve ejaculation. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported strength or force of ejaculation as measured by MSHQ | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 8 will be reviewed from the ejaculation scale. "In the last month, how would you rate the strength or force of your ejaculation?" Measured as (5 = as strong as it always was, 4 = a little less strong than it used to be, 3 = somewhat less strong then it used to be, 2 = much less strong than it used to be, 1 = very much less strong than it used to be, 0= could not ejaculate). A higher score indicates a higher ability to achieve a forceful ejaculation. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported volume of semen when ejaculating as reported on the MSHQ. | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 9 will be reviewed from the ejaculation scale. "In the last month, how would you rate the amount or volume of semen when you ejaculate?" Measured as (5 = as much as it always was time, 4 = a little less then it used to be, 3 = somewhat less than it used to be, 2 = much less than it used to be, 1 = very much less than it used to be, 0= could not ejaculate). A higher score indicates a higher ability to produce a greater volume of ejaculate. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported pleasure with ejaculation as measured by the MSHQ. | At baseline and 4 weeks after completing the primary endpoint
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 10 will be reviewed from the ejaculation scale. "Compared to ONE month ago, would you say the physical pleasure you feel when you ejaculate has-" Measured as (5 = increased a lot, 4 = increased moderately, 3 = neither increased nor decreased, 2 = decreased moderately, 1 = decreased a lot, 0= could not ejaculate). A higher score indicates a higher ability report pleasure with ejaculation. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported pain with ejaculation as measured by the MSHQ. | At baseline and 4 weeks after the primary endpoint visit
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. Specifically the score from question 11 will be reviewed from the ejaculation scale. "In the last month, have you experienced any physical pain or discomfort when you ejaculated? Would you say you have…" Measured as (5 = no pain at all, 4 = slight amount of pain or discomfort, 3 = moderate amount of pain or discomfort, 2 = strong amount of pain or discomfort, 1 = extreme amount of pain or discomfort, 0= could not ejaculate). A higher score indicates no pain or less pain with ejaculation. Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported satisfaction with sex life as measured by the MSHQ. | At baseline and 4 weeks after the primary endpoint visit
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. The MSHQ contains 3 domains: Erection scale (3 items), Ejaculation scale (7 items), and Sexual satisfaction scale (6 items). 9 additional items (2 items measuring bothersome linked to erection and ejaculation and 7 items measuring sexual activity and desire).
  Specifically the score from question 14 will be reviewed from the sexual satisfaction scale. "Generally, how satisfied are you with the quality of the sex life you have with your main partner?" Measured as (5 = extremely satisfied, 4 = moderately satisfied, 3 = neither satisfied nor unsatisfied, 2 = moderately unsatisfied, 1 = extremely unsatisfied). Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
Change in subject-reported urge or desire to have sex as measured by the MSHQ. | At baseline and 4 weeks after the primary endpoint visit
  The MSHQ is a validated, self-administered questionnaire which was developed specifically for assessing key aspects of sexual function and satisfaction in the aging male with urogenital health concerns. The MSHQ contains 3 domains: Erection scale (3 items), Ejaculation scale (7 items), and Sexual satisfaction scale (6 items). 9 additional items (2 items measuring bothersome linked to erection and ejaculation and 7 items measuring sexual activity and desire).
  Specifically question 22 will be reviewed, concerning the sexual urges they have felt toward their main partner, and not whether they actually had sex. "In the last month, how often have you felt an urge or desire to have sex with your main partner?" Measured as (5 =all the time, 4 = most of the time, 3 = about half of the time, 2 = less than half of the time, 1 = none of the time). Change from baseline is reported, with a positive number indicating a worsening and a negative number indicating improvement.
The secondary durability objective for this study is to determine whether subjects in the Emsella Chair group continue to have a higher responder rate, compared to the Sham group, as measured by the GRA. | 4 weeks after the primary endpoint visit
  The GRA is a validated single question survey prompting subjects to rank change in symptom severity since the start of therapy on a 7-point scale (1 = markedly worse, 2 = moderately worse, 3 = mildly worse, 4 = same, 5= slightly improved, 6 = moderately improved, 7= markedly improved). A higher score indicates a better outcome.
The secondary safety objective of this study are to determine the safety and tolerability of the Emsella Chair compared to Sham. Safety and tolerability will be assessed in relation to the incidence of adverse events. | Approximately 12 weeks, up to 24
  Adverse event monitoring will occur between start of treatment to the end of study participation, approximately 12 weeks including the last follow-up visit of the blinded portion. Those randomized to the sham treatment will be offered active treatment after the secondary endpoint visit is completed. Those that elect to receive active treatment will be monitored for adverse events through the last follow-up visit, events during this timeframe will be considered active Emsella Chair.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States